CLINICAL TRIAL: NCT04700995
Title: Postoperative Pain After Endodontic Retreatment Using Different Rotary or Reciprocating Instruments: A Randomized, Controlled Clinical Trial
Brief Title: Postoperative Pain After Using NiTi Instruments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Burhan Can Çanakçi, Assistant Professor, Trakya University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TrakyaU 2020/150
Record Dates: First submitted 2021-01-05; First posted 2021-01-08 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Post-Op Complication; Endodontic Inflammation; Endodontically Treated Teeth; Apical Periodontitis
Keywords: non-surgical endodontic retreatment; post operative pain; rotary NiTi instrument; reciprocating NiTi instrument; ProTaper Universal; ProTaper Gold; Hyflex EDM; Reciproc Blue; WaveOne Gold
MeSH Terms: conditions — Postoperative Complications; Pulpitis; Tooth, Nonvital; Periapical Periodontitis; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ProTaper rotary NiTi instruments (Experimental): The ProTaper Universal Retreatment rotary system and ProTaper Gold rotary system were used.
  Interventions: Procedure: NiTi instruments
- Hyflex EDM rotary NiTi instruments (Experimental): Hyflex EDM rotary system was used.
  Interventions: Procedure: NiTi instruments
- Reciproc Blue reciprocating NiTi instruments (Experimental): Reciproc Blue reciprocating system was used.
  Interventions: Procedure: NiTi instruments
- Waveone Gold reciprocating NiTi instruments (Experimental): WaveOne Gold reciprocating system was used.
  Interventions: Procedure: NiTi instruments

INTERVENTIONS:
Procedure: NiTi instruments — Root canal filling removal

SUMMARY:
The aim of this randomized clinical trial was to compare the incidence, intensity and duration of postoperative pain following the removal of root canal obturation materials canals using rotary (ProTaper Universal or Hyflex EDM) or reciprocating file (Reciproc Blue or WaveOne Gold) systems. The null hypothesis tested was that there is no difference in postoperative pain following the retreatment procedure between the four systems used.

DETAILED DESCRIPTION:
Postoperative pain (PP) is not a certain reason for the long term success of root canal treatment. However, PP control is important for patient comfort and satisfaction. Apical extrusion of debris containing dentin, necrotic pulp tissue, microorganisms, and/or irrigation solutions may occur during retreatment procedures which may result in the induction of periapical inflammation, postoperative pain, and delayed periapical healing. All available techniques and instruments are associated with apical extrusion of debris to some degree during the root canal preparation or removal of the obturation materials. The aim of this randomized clinical trial was to compare the incidence, intensity and duration of postoperative pain following the removal of root canal obturation materials canals using rotary or reciprocating file systems.

Patients referred for non-surgical endodontic retreatment were included. Hundred and eighty cases were selected on the basis of the determined inclusion criteria and randomly allocated to four groups (n = 45).

ProTaper Universal group D1, D2 and D3 files were used respectively with a full rotational motion with a endodontic motor until working was reached as recommended by the manufacturer.

Hylex EDM group Hylex EDM files were used with a full rotational motion with a endodontic motor until the working was reached.

Reciproc Blue group R25 files were used with a reciprocating motion using with the "RECIPROC ALL" mode with a slow in-and-out pecking motion, and the amplitude of pecking movements did not exceed 3 mm until the working lenght was reached.

Waveone Gold group Primary files were used with a reciprocating motion using with the "WAVEONE ALL" mode with a slow in-and-out pecking motion, and the amplitude of pecking movements did not exceed 3 mm until the working was reached.

Assessment of postoperative pain Before participation, all patients had read and signed an informed consent form., all patients were given a pain report form on which they would report their preoperative level of pain.

Before beginning of treatment, the clinician filled in an example of pain report with each patient to confirm that they understood the instructions.

The degree of the postoperative pain was measured using an 11-level numeric rating scale (NRS) at 24, 48, and 72 h following the retreatment. The NRS is a segmented numeric version of the visual analog scale (VAS) and consists of successive numbers from 0 to 10 on a horizontal line. The respondent selects a number that best represents the intensity of his pain. Number "0" represents "no pain" whereas number "10" represents "the worst pain imaginable".

Patients were asked to fill out forms at relevant times in accordance with the instructions given.

An analgesic tablet (400 mg Ibuprofen) was prescribed to take an in case of severe pain, at 6-h intervals. Also they were requested to record the number of analgesic pills consumed each day. The forms were collected on the 4th day following the retreatment. Also a phone call was made every day for 3 days to obtain information on the postoperative pain and the frequency of analgesic intake. The patients were asked to call the contact number on the form if they encountered severe pain or if they needed to ask any questions regarding the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy patient who has a failed root canal treatment.
* Asymptomatic single rooted teeth that had an initial root canal filling diagnosed with chronic apical periodontitis.
* Patients agreed to parcitipate in the study

Exclusion Criteria:

* Overfilled teeth,
* teeth with intraradicular posts,
* existence of a sinus tract,
* consumption of antibiotics or analgesics within one month,
* pregnancy,
* history of trauma,
* traumatic occlusion

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-10 (Actual)

PRIMARY OUTCOMES:
Postoperative pain after removal of gutta-percha using four different NiTi systems. | 24 hours postoperatively
  Pain intensity was evaluated at 24 hours after retreatment procedures. An 11 item numerical rating scale (NSR) was used to assess the pain. The NSR is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of their pain. The number 0 represents "no pain" wheres number 10 represents "pain as bad as someone can imagine". All patients were requested to mark a number corresponding to their average pain.

SECONDARY OUTCOMES:
Postoperative pain after removal of gutta-percha using four different NiTi systems. | 24 to 48 hours postoperatively
  Pain intensity was evaluated at 48 hours after retreatment procedures. An 11 item numerical rating scale (NSR) was used to assess the pain. The NSR is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of their pain. The number 0 represents "no pain" wheres number 10 represents "pain as bad as someone can imagine". All patients were requested to mark a number corresponding to their average pain.

OTHER OUTCOMES:
Postoperative pain after removal of gutta-percha using four different NiTi systems. | 48 to 72 hours postoperatively
  Pain intensity was evaluated at 72 hours after retreatment procedures. An 11 item numerical rating scale (NSR) was used to assess the pain. The NSR is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of their pain. The number 0 represents "no pain" wheres number 10 represents "pain as bad as someone can imagine". All patients were requested to mark a number corresponding to their average pain.

CONTACTS AND LOCATIONS:
Overall Officials: Burhan Çanakçi, Principal Investigator — Trakya University, Faculty of Dentistry; Özgür Er, Study Director — Trakya University, Faculty of Dentistry
Locations (1):
- Burhan Çanakçi, Edirne, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No